CLINICAL TRIAL: NCT00468728
Title: A Double-Blind Study to Compare the Safety and Efficacy of PAR-101 to Vancomycin in Subjects With Clostridium Difficile-Associated Diarrhea (CDAD)
Brief Title: PAR-101/OPT-80 Versus Vancomycin for the Treatment of Clostridium Difficile-Associated Diarrhea (CDAD)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Optimer Pharmaceuticals LLC, a subsidiary of Merck & Co., Inc. (Rahway, New Jersey USA) (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 5119-019; 101.1.C.004 (Other: Optimerpharma Study Number); NCT00427869 (obsolete NCT alias)
Record Dates: First submitted 2007-05-01; First posted 2007-05-03 (Estimated); Results first posted 2011-07-29 (Estimated); Last update posted 2017-04-21 (Actual); Status verified 2017-03

CONDITIONS: Clostridium Infections; Diarrhea
Keywords: CDAD, Clostridium difficile, diarrhea; Clostridium difficile-Associated Diarrhea
MeSH Terms: conditions — Clostridium Infections; Diarrhea | interventions — Vancomycin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator): Vancomycin
  Interventions: Drug: Vancomycin
- 2 (Experimental): PAR-101/OPT-80
  Interventions: Drug: PAR-101/OPT-80

INTERVENTIONS:
Drug: PAR-101/OPT-80 — capsules
  Arms: 2
Drug: Vancomycin — Capsules
  Arms: 1

SUMMARY:
This is a comparative study to investigate the safety and efficacy of PAR-101/OPT-80 (fidaxomicin) versus vancomycin in subjects with Clostridium difficile-associated diarrhea (CDAD).

DETAILED DESCRIPTION:
The primary objective of this pivotal study is to investigate the safety and efficacy of PAR-101/OPT-80 versus vancomycin in subjects with Clostridium difficile-associated diarrhea (CDAD). The cure rates at end of therapy and recurrence rates will be evaluated and compared.

ELIGIBILITY:
Inclusion Criteria:

* Males/females with CDAD
* Females must use adequate contraception
* Signed informed consent

Exclusion Criteria:

* Life-threatening CDAD
* Toxic megacolon
* Pregnant
* Concurrent use of diarrheal agents
* Participation in other trials

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 535 (Actual)
Dates: Start 2006-10-04 (Actual); Primary Completion 2009-12-11 (Actual); Study Completion 2009-12-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dr. Sherwood Gorbach, MD, Study Director — Optimer Pharmaceuticals, Inc.
Locations (116):
- United States (53):
  - Gadsden, Alabama
  - Phoenix, Arizona
  - Hot Springs, Arkansas
  - La Mesa, California
  - Modesto, California
  - Palm Springs, California
  - Rancho Mirage, California
  - San Jose, California
  - Santa Ana, California
  - Vallejo, California
  - Washington D.C., District of Columbia
  - Miami, Florida
  - Port Orange, Florida
  - Sarasota, Florida
  - Marietta, Georgia
  - Savannah, Georgia
  - Idaho Falls, Idaho
  - Chicago, Illinois
  - Maywood, Illinois
  - Indianapolis, Indiana
  - Bowling Green, Kentucky
  - Jena, Louisiana
  - New Orleans, Louisiana
  - Baltimore, Maryland
  - Boston, Massachusetts
  - West Roxbury, Massachusetts
  - Detroit, Michigan
  - Keego Harbor, Michigan
  - Royal Oak, Michigan
  - Minneapolis, Minnesota
  - Tupelo, Mississippi
  - Columbia, Missouri
  - Butte, Montana
  - Cedar Knolls, New Jersey
  - Neptune City, New Jersey
  - The Bronx, New York
  - Charlotte, North Carolina
  - Winston-Salem, North Carolina
  - Fargo, North Dakota
  - Akron, Ohio
  - Amherst, Ohio
  - Cleveland, Ohio
  - Columbus, Ohio
  - Dayton, Ohio
  - Philadelphia, Pennsylvania
  - Pittsburgh, Pennsylvania
  - Charleston, South Carolina
  - Rapid City, South Dakota
  - Sioux Falls, South Dakota
  - San Antonio, Texas
  - Winchester, Virginia
  - Seattle, Washington
  - Charleston, West Virginia
- Belgium (11):
  - Aalst
  - Alast
  - Antwerp
  - Brussels
  - Columbia
  - Ghent
  - Kortrijk
  - Liège
  - Mons
  - Montigny-le-Tilleul
  - Wilrijk
- Canada (9):
  - Calgary, Alberta
  - Edmonton, Alberta
  - Hamilton, Ontario
  - Toronto, Ontario
  - Chicoutimi, Quebec
  - Montreal, Quebec
  - Saint-Jérôme, Quebec
  - Sherbrooke, Quebec
  - Trois-Rivières, Quebec
- France (9):
  - Amiens
  - Caen
  - Clichy
  - Garches
  - Grenoble
  - Lille
  - Tourcoing
  - Tours
  - Valenciennes
- Germany (8):
  - Cologne
  - Düsseldorf
  - Frankfurt
  - Hanover
  - Hofheim am Taunus
  - Lübeck
  - Magdeburg
  - Regensburg
- Italy (5):
  - Busto Arsizio
  - Genova
  - Milan
  - Modena
  - Torino
- Spain (5):
  - Badalona
  - Barcelona
  - Madrid
  - Palma de Mallorca
  - Seville
- Sweden (3):
  - Eskilstuna
  - Gothenburg
  - Örebro
- United Kingdom (13):
  - Great Yarmouth, Norfolk
  - Derriford, Plymouth
  - Barnsley
  - Brighton
  - Cambridge
  - Edinburgh
  - Liege
  - London
  - Nottingham
  - Oxford
  - Oxon
  - Surrey
  - York

IPD SHARING:
Plan to Share IPD: Yes
http://www.merck.com/clinical-trials/pdf/Merck%20Procedure%20on%20Clinical%20Trial%20Data%20Access%20Final_Updated%20July_9_2014.pdf
  http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- [Result] Cornely OA, Crook DW, Esposito R, Poirier A, Somero MS, Weiss K, Sears P, Gorbach S; OPT-80-004 Clinical Study Group. Fidaxomicin versus vancomycin for infection with Clostridium difficile in Europe, Canada, and the USA: a double-blind, non-inferiority, randomised controlled trial. Lancet Infect Dis. 2012 Apr;12(4):281-9. doi: 10.1016/S1473-3099(11)70374-7. Epub 2012 Feb 8. PMID 22321770
- [Derived] D'Agostino RB Sr, Collins SH, Pencina KM, Kean Y, Gorbach S. Risk estimation for recurrent Clostridium difficile infection based on clinical factors. Clin Infect Dis. 2014 May;58(10):1386-93. doi: 10.1093/cid/ciu107. Epub 2014 Mar 5. PMID 24599770
- [Derived] Cornely OA, Miller MA, Fantin B, Mullane K, Kean Y, Gorbach S. Resolution of Clostridium difficile-associated diarrhea in patients with cancer treated with fidaxomicin or vancomycin. J Clin Oncol. 2013 Jul 1;31(19):2493-9. doi: 10.1200/JCO.2012.45.5899. Epub 2013 May 28. PMID 23715579
- [Derived] Cornely OA, Miller MA, Louie TJ, Crook DW, Gorbach SL. Treatment of first recurrence of Clostridium difficile infection: fidaxomicin versus vancomycin. Clin Infect Dis. 2012 Aug;55 Suppl 2(Suppl 2):S154-61. doi: 10.1093/cid/cis462. PMID 22752865
- [Derived] Figueroa I, Johnson S, Sambol SP, Goldstein EJ, Citron DM, Gerding DN. Relapse versus reinfection: recurrent Clostridium difficile infection following treatment with fidaxomicin or vancomycin. Clin Infect Dis. 2012 Aug;55 Suppl 2(Suppl 2):S104-9. doi: 10.1093/cid/cis357. PMID 22752857

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were enrolled from April 2007 to November 2009 by centers in the United States, Canada, France, Spain, Belgium, Germany, United Kingdom, Italy, and Sweden.
Groups:
- Vancomycin: 125 mg administered 4 times daily (q6hr)
- PAR-101/OPT-80: 200 mg administered twice daily (q12hr)
Period: Enrollment
Arm/Group | Vancomycin | PAR-101/OPT-80
Started | 264 | 271
Completed | 260 (1 fidaxomicin subject received vancomycin, 11 subjects didn't take drug) | 264 (1 fidaxomicin subject received vancomycin, 11 subjects didn't take drug)
Not Completed | 4 | 7
Period: Treatment
Arm/Group | Vancomycin | PAR-101/OPT-80
Started | 260 | 264
Completed | 256 | 253
Not Completed | 4 | 11
Not completed — criteria for mITT population | 4 | 11
Period: Follow-up
Arm/Group | Vancomycin | PAR-101/OPT-80
Started | 256 | 253
Completed | 222 | 222
Not Completed | 34 | 31
Not completed — mITT failure | 34 | 31

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Vancomycin | PAR-101/OPT-80 | Total
Number analyzed (Participants) | 256 | 253 | 509
Age, Continuous [Mean (Standard Deviation); unit: years] | 62.7 (18.3) | 64.1 (18.0) | 63.4 (18.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 161 | 149 | 310
  Male | 95 | 104 | 199
Region of Enrollment [Number; unit: participants]
  France | 8 | 11 | 19
  United States | 76 | 74 | 150
  Canada | 82 | 79 | 161
  Spain | 4 | 5 | 9
  Belgium | 20 | 22 | 42
  Germany | 19 | 18 | 37
  United Kingdom | 27 | 26 | 53
  Italy | 13 | 14 | 27
  Sweden | 7 | 4 | 11

OUTCOME MEASURES:

1. Primary Outcome: Cure Rate at End of Therapy
Description: Percentage of subjects with 3 or fewer unformed stools for 2 consecutive days and maintained through the end of therapy, and the subject no longer needed specific anti-Clostridium antibacterial treatment after completion of the course of study medication.
Time Frame: Study day 10 (+/- 2 days)
Population: Analysis data is modified intent to treat (mITT) population. The mITT population consists of subjects that had CDAD confirmed by >3 unformed bowel movements in the 24 hours prior to randomization and a positive toxin assay and received at least one dose of study medication.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Vancomycin | PAR-101/OPT-80
Number analyzed (Participants) | 256 | 253
Percentage of Participants | 86.7 [82.0 to 90.4] | 87.7 [83.1 to 91.2]
Statistical Analysis 1: Comparison: Vancomycin vs PAR-101/OPT-80; H0: C(OPT-80) - C(VAN) <= -10% Power calculation is based on cure rate of 85% in both treatment groups, non-inferiority margin of 10%, 2.5% (1-sided) type I error rate with approximately 90% power gives a total of 530 subjects; Test type: Non-Inferiority or Equivalence — The point estimate of the difference and the 2-sided 95% confidence interval (CI) for the difference between treatment groups were computed. If the lower limit of the CI was greater than -10%, the clinical non-inferiority of fidaxomicin was demonstrated. CIs for the difference of cure rates were calculated using the method recommended by Agresti and Caffo; Risk Difference (RD) = 1.0, 95% CI 2-sided [-4.8 to 6.8]

2. Secondary Outcome: Recurrence
Description: Percentage of subjects with the re-establishment of diarrhea to an extent(based on frequency of passed unformed stools) that was greater than that noted on the last day of study medication, and the demonstration of either toxin A or B or both of C. difficile, and retreatment with CDI anti-infective therapy was needed.
Time Frame: Study days 11-40
Population: The analysis population is mITT, for subjects who met the primary endpoint of cure, was analyzed for the recurrence rates of diarrhea up to the Poststudy Visit.
Measure: Number; unit: Percentage of Participants
Groups:
- Vancomycin: 125 mg administered 4 times daily
- PAR-101/OPT-80: 200 mg administered twice daily
Arm/Group | Vancomycin | PAR-101/OPT-80
Number analyzed (Participants) | 222 | 222
Percentage of Participants | 27.0 | 12.6
Statistical Analysis 1: Comparison: Vancomycin vs PAR-101/OPT-80; Test type: Superiority or Other; p < 0.001, Chi-squared; Risk Difference (RD) = -14.4, 95% CI 2-sided [-21.6 to -7.0]

3. Secondary Outcome: Global Cure
Description: Achieving a cure response at end of treatment and not having a recurrence at any time up to the post-study visit.
Time Frame: End of Study
Population: The analysis population is mITT, subjects that achieved a cure response at end of treatment and not having a recurrence at any time up to the Post-study visit.
Measure: Number; unit: Percentage of Participants
Arm/Group | Vancomycin | PAR-101/OPT-80
Number analyzed (Participants) | 256 | 253
Percentage of Participants | 63.3 | 76.7
Statistical Analysis 1: Comparison: Vancomycin vs PAR-101/OPT-80; Test type: Superiority or Other; p = 0.001, Chi-squared; Risk Difference (RD) = 13.4, 95% CI [5.4 to 21.1]

ADVERSE EVENTS:
Time Frame: From Informed consent to 7-days following the last dose of study drug or until the last protocol-specified study visit, whichever occured later.
Arm/Group | Vancomycin | PAR-101/OPT-80
Serious Adverse Events (participants affected / at risk) | 58/260 | 70/264
Other Adverse Events (participants affected / at risk) | 177/260 | 186/264
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Vancomycin (N=260) | PAR-101/OPT-80 (N=264)
ANAEMIA (Blood and lymphatic system disorders) | 1 | 0
LYMPHOPENIA (Blood and lymphatic system disorders) | 1 | 2
LEUKOPENIA (Blood and lymphatic system disorders) | 0 | 3
NEUTROPENIA (Blood and lymphatic system disorders) | 0 | 4
THROMBOCYTOPENIA (Blood and lymphatic system disorders) | 0 | 3
CARDIO-RESPIRATORY ARREST (Cardiac disorders) | 2 | 0
CARDIAC FAILURE CONGESTIVE (Cardiac disorders) | 1 | 1
TORSADE DE POINTES (Cardiac disorders) | 1 | 0
ATRIAL FIBRILLATION (Cardiac disorders) | 0 | 1
MYOCARDIAL INFARCTION (Cardiac disorders) | 0 | 4
SMALL INTESTINAL OBSTRUCTION (Gastrointestinal disorders) | 3 | 0
VOMITING (Gastrointestinal disorders) | 3 | 1
ABDOMINAL REBOUND TENDERNESS (Gastrointestinal disorders) | 1 | 0
ANAL FISSURE (Gastrointestinal disorders) | 1 | 0
DIARRHOEA (Gastrointestinal disorders) | 1 | 1
FAECAL VOMITING (Gastrointestinal disorders) | 1 | 0
ILEUS PARALYTIC (Gastrointestinal disorders) | 1 | 0
INTESTINAL OBSTRUCTION (Gastrointestinal disorders) | 1 | 3
OESOPHAGEAL VARICES HAEMORRHAGE (Gastrointestinal disorders) | 1 | 0
UPPER GASTROINTESTINAL HAEMORRHAGE (Gastrointestinal disorders) | 1 | 0
ABDOMINAL PAIN (Gastrointestinal disorders) | 0 | 3
COLITIS (Gastrointestinal disorders) | 0 | 1
CROHN'S DISEASE (Gastrointestinal disorders) | 0 | 1
DIARRHOEA HAEMORRHAGIC (Gastrointestinal disorders) | 0 | 2
FEMORAL HERNIA (Gastrointestinal disorders) | 0 | 1
GASTROINTESTINAL PERFORATION (Gastrointestinal disorders) | 0 | 1
MEGACOLON (Gastrointestinal disorders) | 0 | 1
NAUSEA (Gastrointestinal disorders) | 0 | 1
PERITONITIS (Gastrointestinal disorders) | 0 | 1
MULTI-ORGAN FAILURE (General disorders) | 2 | 0
PYREXIA (General disorders) | 2 | 2
EUTHANASIA (General disorders) | 1 | 0
CHEST PAIN (General disorders) | 0 | 1
HEPATIC CIRRHOSIS (Hepatobiliary disorders) | 1 | 0
HYPERBILIRUBINAEMIA (Hepatobiliary disorders) | 1 | 0
CHOLESTASIS (Hepatobiliary disorders) | 0 | 1
PNEUMONIA (Infections and infestations) | 5 | 4
CLOSTRIDIUM DIFFICILE COLITIS (Infections and infestations) | 3 | 5
CLOSTRIDIAL INFECTION (Infections and infestations) | 2 | 1
ESCHERICHIA SEPSIS (Infections and infestations) | 2 | 0
SEPSIS (Infections and infestations) | 2 | 4
UROSEPSIS (Infections and infestations) | 2 | 1
CLOSTRIDIUM DIFFICILE SEPSIS (Infections and infestations) | 1 | 0
ENDOCARDITIS (Infections and infestations) | 1 | 0
INFLUENZA (Infections and infestations) | 1 | 0
LOCALISED INFECTION (Infections and infestations) | 1 | 0
OSTEOMYELITIS (Infections and infestations) | 1 | 0
PNEUMONIA FUNGAL (Infections and infestations) | 1 | 0
SEPTIC SHOCK (Infections and infestations) | 1 | 0
STAPHYLOCOCCAL SEPSIS (Infections and infestations) | 1 | 0
SYSTEMIC CANDIDA (Infections and infestations) | 1 | 0
BETA HAEMOLYTIC STREPTOCOCCAL INFECTION (Infections and infestations) | 0 | 1
BRONCHOPULMONARY ASPERGILLOSIS (Infections and infestations) | 0 | 1
EAR INFECTION (Infections and infestations) | 0 | 1
ERYSIPELAS (Infections and infestations) | 0 | 1
LIVER ABSCESS (Infections and infestations) | 0 | 1
NEUTROPENIC SEPSIS (Infections and infestations) | 0 | 1
PNEUMONIA KLEBSIELLA (Infections and infestations) | 0 | 1
STAPHYLOCOCCAL INFECTION (Infections and infestations) | 0 | 1
SUBACUTE ENDOCARDITIS (Infections and infestations) | 0 | 1
URINARY TRACT INFECTION (Infections and infestations) | 0 | 1
HIP FRACTURE (Injury, poisoning and procedural complications) | 1 | 1
INJURY (Injury, poisoning and procedural complications) | 1 | 0
FALL (Injury, poisoning and procedural complications) | 0 | 1
FEMORAL NECK FRACTURE (Injury, poisoning and procedural complications) | 0 | 1
JOINT DISLOCATION (Injury, poisoning and procedural complications) | 0 | 1
ALANINE AMINOTRANSFERASE INCREASED (Investigations) | 2 | 1
ASPARTATE AMINOTRANSFERASE INCREASED (Investigations) | 1 | 0
BLOOD GLUCOSE INCREASED (Investigations) | 1 | 0
BLOOD PHOSPHORUS ABNORMAL (Investigations) | 1 | 0
BLOOD POTASSIUM DECREASED (Investigations) | 1 | 0
ELECTROCARDIOGRAM QT PROLONGED (Investigations) | 1 | 0
HEPATIC ENZYME INCREASED (Investigations) | 1 | 1
LIPASE INCREASED (Investigations) | 1 | 0
LIVER FUNCTION TEST ABNORMAL (Investigations) | 1 | 1
LYMPHOCYTE COUNT ABNORMAL (Investigations) | 1 | 0
BLOOD ALKALINE PHOSPHATASE INCREASED (Investigations) | 0 | 1
BLOOD BICARBONATE DECREASED (Investigations) | 0 | 1
BLOOD URIC ACID INCREASED (Investigations) | 0 | 2
LYMPHOCYTE COUNT DECREASED (Investigations) | 0 | 3
NEUTROPHIL COUNT DECREASED (Investigations) | 0 | 1
HYPERGLYCAEMIA (Metabolism and nutrition disorders) | 3 | 2
HYPERURICAEMIA (Metabolism and nutrition disorders) | 2 | 1
HYPOKALAEMIA (Metabolism and nutrition disorders) | 2 | 2
DEHYDRATION (Metabolism and nutrition disorders) | 1 | 2
HYPERKALAEMIA (Metabolism and nutrition disorders) | 1 | 3
MALNUTRITION (Metabolism and nutrition disorders) | 1 | 0
HYPONATRAEMIA (Metabolism and nutrition disorders) | 0 | 4
HYPOPHOSPHATAEMIA (Metabolism and nutrition disorders) | 0 | 2
METABOLIC ACIDOSIS (Metabolism and nutrition disorders) | 0 | 1
LUNG NEOPLASM MALIGNANT (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
LYMPHATIC SYSTEM NEOPLASM (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
T-CELL LYMPHOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
COLON CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
GALLBLADDER CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
METASTASIS (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
CEREBRAL INFARCTION (Nervous system disorders) | 1 | 0
SYNCOPE (Nervous system disorders) | 0 | 1
ALCOHOLISM (Psychiatric disorders) | 1 | 0
HALLUCINATION (Psychiatric disorders) | 0 | 1
RENAL FAILURE ACUTE (Renal and urinary disorders) | 2 | 0
RENAL FAILURE (Renal and urinary disorders) | 1 | 3
NEPHROLITHIASIS (Renal and urinary disorders) | 0 | 1
RENAL IMPAIRMENT (Renal and urinary disorders) | 0 | 1
URINARY RETENTION (Renal and urinary disorders) | 0 | 1
PROSTATITIS (Reproductive system and breast disorders) | 0 | 1
RESPIRATORY FAILURE (Respiratory, thoracic and mediastinal disorders) | 3 | 3
ACUTE RESPIRATORY FAILURE (Respiratory, thoracic and mediastinal disorders) | 2 | 0
PULMONARY OEDEMA (Respiratory, thoracic and mediastinal disorders) | 2 | 1
EPISTAXIS (Respiratory, thoracic and mediastinal disorders) | 1 | 0
PLEURAL EFFUSION (Respiratory, thoracic and mediastinal disorders) | 1 | 1
PNEUMONIA ASPIRATION (Respiratory, thoracic and mediastinal disorders) | 1 | 0
TACHYPNOEA (Respiratory, thoracic and mediastinal disorders) | 1 | 1
ACUTE PULMONARY OEDEMA (Respiratory, thoracic and mediastinal disorders) | 0 | 1
CHRONIC OBSTRUCTIVE PULMONARY DISEASE (Respiratory, thoracic and mediastinal disorders) | 0 | 1
HYPOXIA (Respiratory, thoracic and mediastinal disorders) | 0 | 1
RESPIRATORY ARREST (Respiratory, thoracic and mediastinal disorders) | 0 | 1
RESPIRATORY DISTRESS (Respiratory, thoracic and mediastinal disorders) | 0 | 2
HYPOTENSION (Vascular disorders) | 1 | 0
HYPERTENSIVE CRISIS (Vascular disorders) | 0 | 1
PERIPHERAL ARTERIAL OCCLUSIVE DISEASE (Vascular disorders) | 0 | 1
PERIPHERAL EMBOLISM (Vascular disorders) | 0 | 1
PERIPHERAL ISCHAEMIA (Vascular disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Vancomycin (N=260) | PAR-101/OPT-80 (N=264)
NAUSEA (Gastrointestinal disorders) | 30 | 25
VOMITING (Gastrointestinal disorders) | 20 | 16
DIARRHOEA (Gastrointestinal disorders) | 14 | 8
ABDOMINAL PAIN (Gastrointestinal disorders) | 11 | 23
ABDOMINAL PAIN UPPER (Gastrointestinal disorders) | 9 | 3
CONSTIPATION (Gastrointestinal disorders) | 6 | 11
DYSPEPSIA (Gastrointestinal disorders) | 6 | 2
ABDOMINAL DISTENSION (Gastrointestinal disorders) | 5 | 9
FLATULENCE (Gastrointestinal disorders) | 3 | 6
FATIGUE (General disorders) | 12 | 9
PYREXIA (General disorders) | 10 | 6
OEDEMA PERIPHERAL (General disorders) | 7 | 4
PNEUMONIA (Infections and infestations) | 8 | 6
URINARY TRACT INFECTION (Infections and infestations) | 5 | 6
CLOSTRIDIUM DIFFICILE COLITIS (Infections and infestations) | 3 | 6
SEPSIS (Infections and infestations) | 2 | 6
ELECTROCARDIOGRAM QT PROLONGED (Investigations) | 3 | 7
HYPOKALAEMIA (Metabolism and nutrition disorders) | 11 | 18
HYPERKALAEMIA (Metabolism and nutrition disorders) | 4 | 6
BACK PAIN (Musculoskeletal and connective tissue disorders) | 7 | 3
PAIN IN EXTREMITY (Musculoskeletal and connective tissue disorders) | 1 | 6
HEADACHE (Nervous system disorders) | 11 | 15
DIZZINESS (Nervous system disorders) | 7 | 3
INSOMNIA (Psychiatric disorders) | 5 | 7
COUGH (Respiratory, thoracic and mediastinal disorders) | 2 | 7
PRURITUS (Skin and subcutaneous tissue disorders) | 8 (8) | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less